CLINICAL TRIAL: NCT06747806
Title: Biobank of Blood and Tissue Samples From Patients Undergoing Cardiac Surgery
Brief Title: Biobank Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB20-1974
Record Dates: First submitted 2024-11-22; First posted 2024-12-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who undergo cardiac surgery and procedures: Patients who undergo cardiac surgery and procedures will have tissue specimens that are removed during surgery and collected blood samples of 5 mL.
  Interventions: Procedure: Cardiac Surgery and Procedures

INTERVENTIONS:
Procedure: Cardiac Surgery and Procedures — To assess blood and tissue biomarkers of patients undergoing cardiac surgery

SUMMARY:
Treatment strategies for cardiac surgery patients have been evolving significantly for the last decade. While clinical outcomes have been improving, there are still significant areas unexplored in these patients. Cardiac surgery, or cardiovascular surgery, is surgery on the heart or great vessels performed by cardiac surgeons. It is often used to treat complications of ischemic heart disease (for example, with coronary artery bypass grafting); to correct congenital heart disease; or to treat valvular heart disease from various causes, including endocarditis, rheumatic heart disease, and atherosclerosis.

Biobanking is a fundamental process required in the better understanding of human diseases together with their underlying mechanisms. Biobanking refers to the process by which samples of bodily fluid or tissue are collected for research use to improve the understanding of health and disease. For this study, the investigator's objective is to acquire elucidation in disease etiology, translation, and advancing public health by evaluating blood and tissue results of those with cardiac disease undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo cardiac surgery at Advocate Children's Hospital (ACH)& University of Chicago Medical Center (UCMC) by the ACH & UC Cardiothoracic Surgery Research team who are pediatric neonates and up.
* Patients will only be English speaking.

Exclusion Criteria:

* Vulnerable Subjects/Subject Capacity to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who undergo cardiac surgery at Advocate Children's Hospital (ACH)& University of Chicago Medical Center (UCMC)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of the elucidation in disease etiology from evaluating blood and tissue results | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To acquire elucidation in disease etiology health by evaluating blood and tissue results of those with cardiac disease undergoing cardiac surgery.
Concentration of the elucidation in disease translation from evaluating blood and tissue results | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To acquire elucidation in disease translational health by evaluating blood and tissue results of those with cardiac disease undergoing cardiac surgery.
Concentration of the elucidation in advancing public health by evaluating blood and tissue results | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To acquire elucidation in advancing public health by evaluating blood and tissue results of those with cardiac disease undergoing cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Valluvan Jeevanandam, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Hyde Park, Illinois, United States